CLINICAL TRIAL: NCT01538823
Title: Urine Proteome of Surgical Patients and Healthy Volunteers.
Acronym: UP
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201202051
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Renal Cell Cancer
Keywords: Surgery, Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Group 1: Enrollment of surgical patients at Barnes Jewish Hospital (BJH) with a presumptive diagnosis of RCC and planned nephrectomy or partial nephrectomy.
- Group 2: Surgical patients at BJH with non urological cancers
- Group 3: Surgical patients at BJH with a presumptive diagnosis of RCC and planned nephrectomy or partial nephrectomy
- Group 4: Surgical patients at BJH with non urological cancers
- Group 5: Healthy volunteers with no history of cancer or renal disease
- Group 6: Patients at BJH/Washington University School of Medicine under post procedure surveillance for RCC recurrence and patients under treatment for metastatic disease.
- Group 7: Patients with a presumptive diagnosis of bladder cancer or prostate cancer

SUMMARY:
The purpose of this study is to define early urinary biomarkers for diagnosis and prognosis of Renal Cell Carcinoma (RCC) with subsequent development of reliable, cost-effective, screening techniques.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Planned procedure with presumptive diagnosis of RCC, bladder or prostate cancer OR control patient undergoing non-urological surgery OR normal healthy volunteer OR post surgical patient with a diagnosis of RCC and under surveillance for reoccurrence of RCC or treatment of metastatic RCC
* Signed, informed consent

Exclusion Criteria:

* Patients on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to have full or partial kidney removal surgery (possibly because of kidney cancer).
  Patients scheduled to have a procedure because you may have bladder or prostate cancer.
  Patients scheduled to have some other type of surgery (non-urological). Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2012-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
evaluation of novel bio markers | 5 years
  The overall objective of our study is to find and evaluate additional novel biomarkers, predictive of disease, that are present and measurable in whole urine of patients undergoing surgery for renal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Morrissey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Hu R, Gupta R, Wang Z, Wang C, Sun H, Singamaneni S, Kharasch ED, Morrissey JJ. Bioplasmonic paper-based assay for perilipin-2 non-invasively detects renal cancer. Kidney Int. 2019 Dec;96(6):1417-1421. doi: 10.1016/j.kint.2019.08.020. Epub 2019 Sep 3. PMID 31668633